CLINICAL TRIAL: NCT02642913
Title: A Multicenter Phase I/II Study of Enzalutamide With and Without Sorafenib in Advanced Hepatocellular Carcinoma Patients
Brief Title: Study of Enzalutamide With and Without Sorafenib in Advanced Hepatocellular Carcinoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry); Mayo Clinic (Other); University of California, San Francisco (Other); University of Southern California (Other); Washington University School of Medicine (Other); Roswell Park Cancer Institute (Other); National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-279
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Enzalutamide; Sorafenib; 15-279
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — enzalutamide; Sorafenib

ARMS (2):
- Enzalutamide without Sorafenib (Experimental): Will get enzalutamide, at the dose approved by the FDA for prostate cancer. If this dose has serious side effects, a lower dose will be given to new patients as they take part in the study. At the end of this part of the study, the recommended dose of enzalutamide will be set for all patients on this study. More patients will then be treated with this dose.
  Interventions: Drug: Enzalutamide
- Enzalutamide with Sorafenib (Experimental): Will get enzalutamide and sorafenib. The first group of patients will get the recommended dose of enzalutamide with sorafenib by mouth either once or twice daily. The dose of sorafenib you receive will depend on when the patient starts the study. At the beginning of the study, patients will be treated with a lower dose of sorafenib. If this dose does not have serious side effects, a higher dose will be given to new patients as they take part in the study.
  Interventions: Drug: Enzalutamide; Drug: Enzalutamide with Sorafenib

INTERVENTIONS:
Drug: Enzalutamide
Drug: Enzalutamide with Sorafenib
  Arms: Enzalutamide with Sorafenib

SUMMARY:
The purpose of this study is to test the safety of enzalutamide with or without sorafenib at different doses. Enzalutamide is approved by the Food and Drug Administration (FDA) for the treatment of advanced prostate cancer. Enzalutamide blocks a protein called the androgen receptor. Experiments on liver cancer cells and animal models show that blocking the androgen receptor causes liver cancer to stop growing. Enzalutamide has not been approved to treat liver cancer. The investigators want to see if enzalutamide is safe for patients with liver cancer who have had their tumors grow on sorafenib. The investigators also want to see how safe and effective sorafenib and enzalutamide are for liver cancer patients that have never been treated with sorafenib. This is the first time enzalutamide and sorafenib are being used together. This treatment may not help treat the participant's cancer.

DETAILED DESCRIPTION:
This is a multicenter, open label, phase I/II study of enzalutamide with or without sorafenib to define the safety, MTD, and pharmacokinetic parameters of each regimen in advanced HCC patients.

The study will have 4 parts as indicated in the Study Schema, an enzalutamide dose escalation (Part 1A), a sorafenib and enzalutamide dose escalation (Part 1B), and dose expansion cohorts for the Part 1A and Part 1B MTDs (Part 2). Dose escalation will occur using a standard 3 + 3 design and is described in Section 4.2.1. For Part 2, the enzalutamide expansion cohort (Part 2A), will enroll 10 patients and is exploratory in nature; however, it will allow for acquisition of additional PK sampling at the MTD, for determination of safety and efficacy. The MTD sorafenib and enzalutamide combination expansion (Part 2B) will be designed using a Simon minimax design to formally evaluate the 4-month PFS.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of HCC reviewed and confirmed at per the local standard of care.
* Advanced unresectable or metastatic disease
* Measurable disease as defined by RECIST version 1.1
* Tissue available for the evaluation of AR by IHC on pretreatment HCC samples. If tissue is not available, a pretreatment biopsy will not be necessary for eligibility
* Age ≥ 18 years-old
* ECOG performance status ≤ 2
* Child-Pugh category A
* Adequate hepatic function defined by:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5.0 x upper limit of normal (ULN)
  * Total Bilirubin ≤ 1.5 x ULN
* Adequate hematologic function defined by:

  * Absolute neutrophil count (ANC) ≥ 1200/mm3 (≥ 1.2 x 10^9/L)
  * Platelets ≥ 75,000/mm3 (≥ 75 x 10^9/L)
  * Hemoglobin ≥ 8 g/dL (≥ 80 g/L)
* Adequate renal function defined by:

  * Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 40 mL/min (using the Cockcroft-Gault equation)
* Patients must be on antiviral therapy per the local standard of care if active or occult hepatitis B (HBV) infection.
* Patients with active hepatitis C (HCV) may not be antiviral therapy.
* Patients with a history of hypertension should be well controlled (BP ≤ 140/90) on a regimen of antihypertensive therapy.
* Gastrointestinal disorders in the opinion of the treating physician that would impair absorption.
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study.
* Patients with history of liver transplantation may be eligible for the dose expansion cohorts (Parts 2A and 2B) of this study provided all eligibility criteria are met and provided the subject has not had any episodes of acute rejection or serious opportunistic infection within 3 months from enrollment.
* Female subjects of childbearing potential must not be pregnant or lactating at screening.
* Participants must be capable of understanding and complying with the protocol requirements and signing informed consent.

  * Certain immunosuppressive agents such as tacrolimus and sirolimus are prohibited due to drug interaction risk thus liver transplant patients who require these medications for immunosuppression are not eligible.
  * Patients receiving everolimus at immunosuppressive dosages are eligible since the everolimus doses used are lower than standard anti-neoplastic dosages and this agent does not demonstrate anti-cancer activity in HCC. Everolimus does not interact adversely like other immunosuppressive agents.

Exclusion Criteria:

* Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma
* For patients who will receive enzalutamide monotherapy, failure or intolerance of prior sorafenib is required for enrollment. For patients who will receive combination therapy, prior sorafenib is excluded.
* Patients may not have received cytotoxic, biologic or small molecule kinase inhibitor systemic therapy f or at least 3 weeks prior to the first dose of study treatment.
* Patients must not have received prior regional therapy such as ablation, embolization, or radiation therapy for at least 2 weeks prior to the first dose of study treatment. Patients who receive such therapy should have evidence of radiologic progression at this site or other progressing measurable disease.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 3 months before study enrollment. Eligible subjects must be without corticosteroid treatment at the time of study enrollment.
* History of seizure including febrile seizure or any condition that may predispose to seizure (e.g., prior stroke, brain arteriovenous malformation, head trauma with loss of consciousness requiring hospitalization). Also, current or prior treatment with antiepileptic medications for the treatment of seizures or history of loss of consciousness or transient ischemic attack within 12 months of enrollment.
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within six months prior to Screening;
  * Uncontrolled angina within three months prior to Screening;
  * Congestive heart failure NYHA class 3 or 4, or subjects with history of congestive heart
  * failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or MUGA scan
  * performed within 3 months results in a left ventricular ejection fraction that is ≥ 45%;
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
* Anticoagulation with warfarin
* Inability to swallow tablets
* Subjects with history of another primary cancer, with the exception of:

  * curatively resected non-melanoma skin cancer;
  * curatively treated cervical carcinoma in situ;
  * other primary solid tumor with no known active disease present in the opinion of the investigator will not affect patient outcome in the setting of current HCC.
* Patients who are on strong inhibitors of CYP2C8, strong or moderate inducers of CY3A4 and CYP2C8 should discontinue these medications 2 weeks prior to the start of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 4 months
  survival is defined as the time from the initiation of study treatment to HCC radiographic progression or death. Four month PFS is defined as the proportion of patients alive and progression free at 4 months. Patients that come out of study before evaluation of the 4 month endpoint without documented progression will be considered as events for the primary endpoint of 4 month PFS. Progression will be by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: James Harding, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of California San Francisco, San Francisco, California
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/